CLINICAL TRIAL: NCT01196715
Title: REGIME: A Randomised Controlled Trial of Prolonged Treatment With Darbepoetin Alpha, With or Without Recombinant Human Granulocyte Colony Stimulating Factor, Versus Best Supportive Care in Patients With Low-risk Myelodysplastic Syndromes (MDS).
Brief Title: Comparison Study of Standard Care Against Combination of Growth Factors Agents for Low-risk Myelodysplastic Syndromes
Acronym: REGIME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Cancer Research UK (Other); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: MDS201001; 2009-017462-23 (EudraCT Number); CRUK/08/009 (Other Grant/Funding Number: CR-UK)
Record Dates: First submitted 2010-07-26; First posted 2010-09-08 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Myelodysplastic Syndrome
Keywords: Quality of Life; Erythroid response; disease progression; survival; Overall erythroid response at 24 weeks; Quality of life at 24 weeks; Quality of life at 12, 36 and 52 weeks; Overall erythroid response at 12 and 52 weeks; Incidence of disease progression; Overall Survival
MeSH Terms: conditions — Myelodysplastic Syndromes; Disease Progression | interventions — Darbepoetin alfa; Filgrastim; Erythrocyte Transfusion; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Darbepoetin Alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alpha
- G-CSF (Active Comparator)
  Interventions: Drug: Filgrastim
- Best Supportive Care (Active Comparator): Red cell transfusion support to achieve a predicted post-transfusion haemoglobin of 11.0 to 12.0 g/dl at a quantity and frequency such that the minimum haemoglobin is never below 8.0 g/dl
  Interventions: Procedure: Blood Red Cell Transfusion

INTERVENTIONS:
Drug: Darbepoetin alpha — Aranesp 500 mcg vials once every 2 weeks.
  Other Names: Aranesp
  Arms: Darbepoetin Alfa
Drug: Filgrastim — 300 mcg vials twice a week, 3-4 days apart
  Other Names: Neupogen
  Arms: G-CSF
Procedure: Blood Red Cell Transfusion — Red cell transfusion support to achieve a predicted post-transfusion haemoglobin of 11.0 to 12.0 g/dl at a quantity and frequency such that the minimum haemoglobin is never below 8.0 g/dl or such that the patient is never excessively symptomatic, according to local transfusion guidelines/policy.
  Other Names: Blood transfusion.
  Arms: Best Supportive Care

SUMMARY:
REGIME is comparing two treatments, with Darbepoetin Alpha (DA) and Filgrastim (Granulocyte Colony Stimulating Factor, G-CSF), to the standard treatment for Myelodysplastic Syndrome (MDS).

After giving Informed Consent patients will undergo a number of tests to confirm eligibility. Once eligibility is confirmed patients will be randomly assigned to one of the three treatments group: A: Darbepoetin Alpha (DA), B: Darbepoetin Alpha and Filgrastim (DA+G-CSF), C: Blood transfusion only. Patients will be required to attend the clinic once a month for 24 weeks. After 24 weeks if a patient has reacted favorably to the treatment they may continue on the treatment regime up to 52 weeks. After week 24 all patients will be required to attend the clinic twice more, at week 36 and 52.

Patients will be followed for a further 5 years to record loss of response, transformation to Acute Myeloid Leukaemia and/or Refractory Anemia with Excess Blasts and death.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged over 18 years, (no upper age limit)
2. ECOG performance status 0-2
3. Life expectancy more than 6 months
4. A confirmed diagnosis of MDS - WHO type:

   * refractory anaemia (RA)
   * hypoplastic RA ineligible for/or failed immunosuppressive therapy (ALG, cyclosporine)
   * refractory anaemia with ring sideroblasts (RARS)
   * refractory cytopenia with multilineage dysplasia
   * myelodysplastic syndrome unclassifiable
5. IPSS low or Int-1, but with BM blasts less than 5%
6. A haemoglobin concentration of less than 10g/dl and/or red cell transfusion dependence
7. Able to understand the implications of participation in the Trial and give written informed consent.

Exclusion Criteria:

1. MDS with bone marrow blasts greater or equal than 5%
2. Myelodysplastic syndrome associated with del(5q)(q31-33) syndrome
3. Chronic myelomonocytic leukaemia (monocytes greater than1.0x109/l)
4. Therapy-related MDS
5. Splenomegaly, with spleen greater or equal than 5 cm from left costal margin
6. Platelets less than 30x109/l
7. Uncorrected haematinic deficiency. Patient deplete to iron, B12 and folate according to local lab ranges
8. Women who are pregnant or lactating.
9. Females of childbearing potential and all males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) for the duration of the study and for up to 3 months after the last dose of study medication. Note: Subjects are not considered of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal
10. Females of childbearing potential must have a negative pregnancy test prior to starting the study.
11. Uncontrolled hypertension, previous venous thromboembolism, or uncontrolled cardiac or pulmonary disease
12. Previous serious adverse events to the study medications or its components
13. Patients who have had previous therapy with ESAs ± G-CSF within 4 weeks of study entry
14. Patients currently receiving experimental therapy, e.g. with thalidomide, or who are participating in another CTIMP.
15. Medical or psychiatric illness, which makes the patient unsuitable or unable to give informed consent.
16. Patients with malignancy requiring active treatment (except hormonal therapy).
17. Patients with a history of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2010-11-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life - To compare the Quality of Life of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | weeks 0
  To compare the Quality of Life of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Haemoglobin response - To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | week 0
  To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Quality of Life - To compare the Quality of Life of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | weeks 12
  To compare the Quality of Life of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Quality of Life - To compare the Quality of Life of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | weeks 24
  To compare the Quality of Life of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Quality of Life - To compare the Quality of Life of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | weeks 36
  To compare the Quality of Life of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Quality of Life - To compare the Quality of Life of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | weeks 52
  To compare the Quality of Life of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Haemoglobine response - To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | week 4
  To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Haemoglobine response - To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | week 8
  To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Haemoglobine response - To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | week 12
  To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Haemoglobine response - To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | week 16
  To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Haemoglobine response - To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | week 20
  To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Haemoglobine response - To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | week 24
  To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Haemoglobine response - To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | week 36
  To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone
Haemoglobine response - To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone | week 52
  To compare the haemoglobin response of low risk Myelodysplastic Syndrome (MDS) patients randomised to receive prolonged treatment with DA alone, DA with G-CSF or best supportive care alone

SECONDARY OUTCOMES:
Utility of prognostic factor and predictive factor assessment | every week
  To assess the utility of prognostic factor and predictive factor assessment, in particular against the predictive model proposed by Hellstrom-Lindberg.
Utility of prognostic factor and predictive factor assessment | week 4
  To assess the utility of prognostic factor and predictive factor assessment, in particular against the predictive model proposed by Hellstrom-Lindberg.
Utility of prognostic factor and predictive factor assessment | week 8
  To assess the utility of prognostic factor and predictive factor assessment, in particular against the predictive model proposed by Hellstrom-Lindberg.
Utility of prognostic factor and predictive factor assessment | week 12
  To assess the utility of prognostic factor and predictive factor assessment, in particular against the predictive model proposed by Hellstrom-Lindberg.
Utility of prognostic factor and predictive factor assessment | week 16
  To assess the utility of prognostic factor and predictive factor assessment, in particular against the predictive model proposed by Hellstrom-Lindberg.
Utility of prognostic factor and predictive factor assessment | week 20
  To assess the utility of prognostic factor and predictive factor assessment, in particular against the predictive model proposed by Hellstrom-Lindberg.
Utility of prognostic factor and predictive factor assessment | week 24
  To assess the utility of prognostic factor and predictive factor assessment, in particular against the predictive model proposed by Hellstrom-Lindberg.
Utility of prognostic factor and predictive factor assessment | week 36
  To assess the utility of prognostic factor and predictive factor assessment, in particular against the predictive model proposed by Hellstrom-Lindberg.
Utility of prognostic factor and predictive factor assessment | week 52
  To assess the utility of prognostic factor and predictive factor assessment, in particular against the predictive model proposed by Hellstrom-Lindberg.

CONTACTS AND LOCATIONS:
Overall Officials: Samir G Agrawal, MRCP FRCPath PhD, Study Director — Barts and The London NHS Trust
Locations (4):
- United Kingdom (4):
  - Birmingham Cancer Research UK Clinical Trial Unit, Birmingham
  - St Bartholomew's Hospital, London
  - CECM Institute of Cancer, London
  - King's College Hospital Haematoloy Laboratory, London